CLINICAL TRIAL: NCT00191620
Title: Randomized Phase II Study of Cisplatin + Gemcitabine Administered Either as Short Infusion or at a Fixed Dose Rate in Non-Small Cell Lung Cancer
Brief Title: Study Comparing Short Infusion Vs. Fixed Dose of Cisplatin + Gemcitabine in Non Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6952; B9E-LA-S350
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

INTERVENTIONS:
Drug: Gemcitabine
Drug: cisplatin

SUMMARY:
The purposes of this study are to determine:

How standard gemcitabine plus cisplatin compares to fixed dose rate of gemcitabine plus cisplatin in the treatment of non-small cell lung cancer.

The safety of standard gemcitabine plus cisplatin and any side effects that might be associated with it as compared to a fixed dose rate of gemcitabine plus cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histologically or cytologically confirmed diagnosis of NSCLC
* Have provided written informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Prior chemotherapy or biologic therapy (approved or experimental) for NSCLC
* Presence of uncontrolled central nervous system (CNS) metastases
* Inability to comply with protocol or study procedures
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2004-03; Study Completion 2006-05

PRIMARY OUTCOMES:
To evaluate the objective response rate (ORR) of the standard (30 minute infusion) versus a fixed dose rate (10 mg/m2/minute) of gemcitabine combined with cisplatin as treatment for advanced NSCLC after treatment completion.

SECONDARY OUTCOMES:
To evaluate progression-free survival of the standard versus a fixed dose rate of gemcitabine combined with cisplatin as treatment for advanced NSCLC.
To evaluate incidence of laboratory and non laboratory adverse events by maximum Common Toxicity Criteria (CTC) toxicity grade and relationship to study drug of the standard versus a fixed dose rate of gemcitabine combined with cisplatin as treatment for

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/ GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/ GMT - 5 hours, EST), or speak with your personal physician, Buenos Aires, Argentina
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/ GMT - 5 hours, EST), or speak with your personal physician, São Paulo, Brazil
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/ GMT - 5 hours, EST), or speak with your personal physician, Santiago, Chile
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/ GMT - 5 hours, EST), or speak with your personal physician, Mexico City, Mexico

REFERENCES:
- [Derived] Pereira JR, Fein L, Del Giglio A, Blajman CR, Richardet E, Schwartsmann G, Orlando M, Hall BJ, West TM, van Kooten M. Gemcitabine administered as a short infusion versus a fixed dose rate in combination with cisplatin for the treatment of patients with advanced non-small cell lung cancer. Lung Cancer. 2007 Oct;58(1):80-7. doi: 10.1016/j.lungcan.2007.05.004. Epub 2007 Jun 22. PMID 17588704